CLINICAL TRIAL: NCT06890611
Title: A Phase 1, Relative Bioavailability Study of Bimagrumab (LY3985863) Test and Reference Materials, and Bimagrumab Test Material Coadministration and Coformulation With Tirzepatide (LY900042), in Healthy Participants
Brief Title: A Study of Bimagrumab Alone (LY3985863) and Bimagrumab With Tirzepatide (LY900042) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27286; J4Z-MC-GIDG (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — bimagrumab; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Bimagrumab Dose 1 Reference Material (Experimental): Participants will receive a single dose of bimagrumab subcutaneously (SC)
  Interventions: Drug: Bimagrumab
- Bimagrumab Dose 1 Test Material + Tirzepatide (Coadministration) (Experimental): Participants will receive a single dose of bimagrumab SC and a single dose of tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Bimagrumab Dose 1 Test Material + Tirzepatide (Coformulation) (Experimental): Participants will receive a single dose of bimagrumab with tirzepatide SC
  Interventions: Drug: Bimagrumab + Tirzepatide Coformulation
- Bimagrumab Dose 2 Test Material + Tirzepatide (Coadministration) (Experimental): Participants will receive bimagrumab SC and tirzepatide SC for 4 weeks
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Bimagrumab Dose 2 Test Material + Tirzepatide (Coformulation) (Experimental): Participants will receive bimagrumab with tirzepatide SC for 4 weeks
  Interventions: Drug: Bimagrumab + Tirzepatide Coformulation

INTERVENTIONS:
Drug: Bimagrumab — Administered SC
  Other Names: LY3985863; BYM338; VER201
  Arms: Bimagrumab Dose 1 Reference Material; Bimagrumab Dose 1 Test Material + Tirzepatide (Coadministration); Bimagrumab Dose 2 Test Material + Tirzepatide (Coadministration)
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Bimagrumab Dose 1 Test Material + Tirzepatide (Coadministration); Bimagrumab Dose 2 Test Material + Tirzepatide (Coadministration)
Drug: Bimagrumab + Tirzepatide Coformulation — Administered SC
  Other Names: LY900042
  Arms: Bimagrumab Dose 1 Test Material + Tirzepatide (Coformulation); Bimagrumab Dose 2 Test Material + Tirzepatide (Coformulation)

SUMMARY:
The main purpose of this study is to evaluate the body concentration of different forms of bimagrumab, administered alone or with tirzepatide. Participation in the study will last about 4.5 months, including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Are considered healthy as determined by medical evaluation including medical history and physical examination
* Have a body mass index (BMI) within the range of 22.0 to 30.0 kilograms per square meter (kg/m2), inclusive

Exclusion Criteria:

* Have current or a history of pancreatitis or hepatitis
* Have a self-reported increase or decrease in body weight, greater than 5 kilograms (kg), within 3 months prior to screening
* Have uncontrolled high blood pressure
* Have taken medications or alternative remedies to promote weight loss within 3 months prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Bimagrumab Test Material | Predose through Week 13
PK: Cmax of Bimagrumab Reference Material | Predose through Week 13
PK: Cmax of Bimagrumab Coadministered with Tirzepatide | Predose through Week 13
PK: Cmax of Tirzepatide Coadministered with Bimagrumab | Predose through Week 16
PK: Cmax of Bimagrumab Coformulated with Tirzepatide | Predose through Week 16
PK: Cmax of Tirzepatide Coformulated with Bimagrumab | Predose through Week 16
PK: Area Under the Curve from Zero to Infinity AUC (AUC(0-∞)) of Bimagrumab Test Material | Predose through Week 13
PK: AUC(0-∞) of Bimagrumab Reference Material | Predose through Week 13
PK: AUC(0-∞) of Bimagrumab Coadministered with Tirzepatide | Predose through Week 13
PK: AUC(0-∞) of Tirzepatide Coadministered with Bimagrumab | Predose through Week 16
PK: AUC(0-∞) of Bimagrumab Coformulated with Tirzepatide | Predose through Week 16
PK: AUC(0-∞) of Tirzepatide Coformulated with Bimagrumab | Predose through Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No